CLINICAL TRIAL: NCT05077397
Title: Is Regional Oxygen Saturation Effective in Predicting Perfusion Parameters and Patient Outcomes in Liver Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Gul Cakmak, Principal investigator, Marmara University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021.03.17
Record Dates: First submitted 2021-09-12; First posted 2021-10-14 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Tissue Injury; Surgery; Absorption; Disorder
Keywords: liver; tissue oxygenation; near infrared spectroscopy; resection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Group 1 (Active Comparator): After the approval of the local ethics committee and written informed consent, 60 ASA I-III patients aged 18-75 years who will undergo liver resection will be included in the study.
  Patients of Group 1 will be monitored by the InSpectra Tissue Spectrometer, StO2, added to standard ASA monitorisation.
  Interventions: Device: StO2
- Group 2 (Active Comparator): After the approval of the local ethics committee and written informed consent, 60 ASA I-III patients aged 18-75 years who will undergo liver resection will be included in the study.
  Patients of Group 2 will be monitored by O3TM Regional Oximeter System, added to standard ASA monitorisation.
  Interventions: Device: O3
- Group 3 (No Intervention): After the approval of the local ethics committee and written informed consent, 60 ASA I-III patients aged 18-75 years who will undergo liver resection will be included in the study.
  Patients of Group 2 will be monitored by standard ASA monitorisation.

INTERVENTIONS:
Device: StO2 — InSpectra Tissue Spectrometer Model 1615 probe (Hutchinson Technology Inc. Hutchinson, MN, USA) probes will be placed on the skin area corresponding to the patients' liver lodge prior to induction of anesthesia. In addition, the probes of both devices will be placed in the renal site on the same side. Basal values will be measured with both devices and StO2 values in the devices will be recorded every 15 minutes. Probes will not be removed during surgery and for 24 hours postoperatively.
  Arms: Group 1
Device: O3 — O3TM Regional Oximeter System (O3 System, Masimo Corporation, Irvine, CA) probes will be placed on the skin area corresponding to the patients' liver lodge prior to induction of anesthesia. In addition, the probes of both devices will be placed in the renal site on the same side. Basal values will be measured with both devices will be recorded every 15 minutes. Probes will not be removed during surgery and for 24 hours postoperatively.
  Arms: Group 2

SUMMARY:
Sudden hypotension, which may develop during liver resection operations performed under general anesthesia, can affect the patient satisfaction at a high rate by causing complications during and after the operation as a result of disrupting the blood supply of the tissues. Although there are standard monitoring methods such as blood pressure, heart rate, and oxygen status that show unwanted hypotension during anesthesia, it is possible to show hypotension in the early period with new generation methods. Although there are many clinical studies proving the effectiveness of these methods, these methods have not yet been included in the standard monitoring methods.

Our prediction in this study is that the development of intraoperative and postoperative complications in patients who will undergo liver surgery, in whom tissue blood flow is monitored with the help of devices, will be less than in patients who are followed up with traditional methods.

If an individual participate in this study, he will not be subjected to any additional procedures other than routine practice during the participant's operation. Before standard general anesthesia for his surgery, heart rate, oxygenation status, blood pressure parameters will be monitored. After the initiation of general anesthesia, the procedures performed in each liver surgery will be applied. In addition, he will be followed by using a probe that allows monitoring of tissue blood flow and reflects a value to the screen, to which it is attached, by simply sticking to his skin.

DETAILED DESCRIPTION:
Intraoperative tissue ischemia correlates with morbidity and mortality in critically ill patients. Therefore, measurement of tissue oxygenation is important in improving postoperative survival. Although values such as pulse oximetry, blood gas analysis, mixed venous oxygen saturation are routinely used to measure systemic oxygenation, regional tissue oxygen saturation measurement has not yet taken place in clinical practice.

The noninvasive measurement of human tissue oxygenation was first performed in 1874 by Karl Von Vierordt, with the detection of the reduction in the amount of infrared radiation passing through an ischemia-affected hand. The first portable oximeter was developed by Glen Milliken in 1942, but the device has only been used as an experimental tool in the aeronautical and physiology laboratory.

Adequate oxygen delivery (QO2) to meet the metabolic needs (VO2) of a tissue undergoing aerobic metabolism is critical for the long-term viability of this tissue. This condition was first described by Adolph Fick. For example, as the metabolic rate increases in peripheral tissues such as skeletal muscle, oxygen delivery will increase, so the amount of oxygen in the venous capillaries decreases and the arteriovenous oxygen difference increases. In addition, according to Fick's law, it is predicted that tissue oxygen delivery will increase with increasing oxygen gradient in microvascular tissue. Various invasive and/or expensive techniques have been developed to understand the balance between oxygen supply and consumption in peripheral tissue according to Fick's law. MR, PET, and arterial/venous catheterization are examples of these.

NIRS (Near Infrared Spectroscopy) Technology NIRS was first used in clinical practice in 1985 to measure cerebral oxygenation in preterm infants. It was developed to measure regional and systemic oxygenation noninvasively and continuously.

Its working principle is based on the measurement by attenuation of light of a certain wavelength (700-1000 nm) by chromophores such as hemoglobin in the sampled tissue by absorbing it in the tissue. The NIRS signal is mainly derived from hemoglobin in the entire vascular space, primarily small vessels (arterioles, capillaries, and venules). As a result, it provides the measurement of tissue hemoglobin or saturation (StO2) by measuring oxy and deoxy hemoglobin in the tissue. NIRS can also assist in estimating the amount of tissue hemoglobin by reflecting either the total tissue hemoglobin (HbT) or the absolute tissue hemoglobin index (THI).

InSpectra Tissue Spectrometer InSpectra Tissue Spectrometer Model 1615 probe (Hutchinson Technology Inc. Hutchinson, MN, USA); It measures the StO2 value by placing it in the area where somatic oxygenation will be measured. In studies with this device, measurements were made mostly in the thenar region, masseter and deltoid muscle.

Basal StO2 values in the thenar region have been shown to be 86%±6% in healthy subjects. In previous studies, the demonstration of peripheral hypoperfusion with the measurement of StO2 in skeletal muscle has been shown as an early indicator of conditions such as shock and hypovolemia. In addition, there are studies in the literature in which morbidity and mortality follow-up by measuring StO2 in critical patient follow-up such as sepsis. It has been shown that StO2 values below 75% are associated with adverse clinical outcomes in septic patients. In some studies conducted with trauma patients, StO2 measurement after the vascular occlusion test was found to be ineffective as an indicator of early hypoperfusion. In major surgeries such as cardiac surgery and colon resection, significant results have been found by monitoring morbidity, mortality, and postoperative complications with peripheral perfusion measurement. In the literature, hepatic StO2 measurement has been made in pediatric cases and experimental studies; There is no study in which somatic oxygenation measurement was performed in liver resection surgeries in adult patients.

O3TM Regional Oximeter System The O3TM Regional Oximeter System (O3 System, Masimo Corporation, Irvine, CA) is a non-invasive oximeter used to measure and monitor regional oxygen saturation (rSO2) in tissue. O3 sensors are used to measure somatic oxygen saturation in adult patients weighing 40 kg or more.

Parameters that can be measured with this device: rSO2, AUC index ( area under the curve), baseline, delta baseline (Δbase), delta SpO2 (ΔSpO2), Delta HHb (ΔHHb), Delta O2Hb (ΔO2Hb), Delta cHb (ΔcHb).

rSO2 is displayed as a percentage and is a measurement of the regional tissue oxygen saturation value in the local tissue at the sensor site.

Delta SpO2 is also displayed as a percentage and is found by calculating the difference between SpO2 and rSO2.

The delta baseline reflects the change of current rSO2 values relative to the rSO2 value initially shown as a percentage. In order to measure this value, basal rSO2 measurement should be made by pressing the "set baseline" button when the device is connected to the patient.

AUC (min-%) measures the time and depth that the patient stays below the user-defined rSO2 low alarm limit (LAL). Time (minutes) refers to the time the patient stays below the LAL rSO2 value. Depth (%) expresses the magnitude of the difference between the patient's rSO2 level and the LAL rSO2. AUC; It increases when the rSO2 value falls below the defined LAL value. AUC has not been studied in the literature yet, and it has been observed in clinical experience that tissue oxygenation becomes critical when the AUC value is around 500.

Delta HHb, Delta O2Hb and Delta cHb; these features are displayed when the head is selected as the sensor region.

Since tissue hypoperfusion may develop especially in the vascular clamp stage of liver resection surgeries, it is thought that the measurement of peripheral tissue oxygenation in standard monitoring may have a positive effect on patient outcomes.

In the present observational study, the investigators will evaluate the effects of hepatic and renal StO2 measurement on early hypoperfusion and postoperative survival in hepatectomy cases, and peripheral tissue oxygen saturation measurement with StO2 InSpectra Tissue Spectrometer Model 1615 probe (Hutchinson Technology Inc. Hutchinson, MN, USA) and O3TM Regional Oximeter System) The investigators aimed to observe by doing it with O3 System, Masimo Corporation, Irvine, CA) devices. The secondary aim of the study is that these values; age, anatomical region, ASA physical condition, whether it will be affected by the vascular clamp duration and its correlation with the risk of developing postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

- patients with ASA I-III physical status

patients between the ages of 18-75

patients who will undergo liver resection

Exclusion Criteria:

- patients with ASA physical status of IV

patients with clinically significant cardiovascular, respiratory, renal or metabolic disease, ischemic cerebrovascular disease

Patients who have BMI >30

Patients who aged >75 years

Patients with intellectual disability

Patients who will have intraoperative surgical complications

Patients who will need for postoperative ventilation

Patients who have methemoglobinemia after intravascular dye injection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-12-16 (Actual); Primary Completion 2022-03-15 (Estimated); Study Completion 2022-03-20 (Estimated)

PRIMARY OUTCOMES:
Hepatic and renal tissue oxygenation | baseline STO2 and O3 measurements at the beginning of the operation
  we will evaluate the effects of hepatic and renal StO2 measurement on early hypoperfusion and postoperative survival in hepatectomy cases, and peripheral tissue oxygen saturation measurement with StO2 InSpectra Tissue Spectrometer Model 1615 probe (Hutchinson Technology Inc. Hutchinson, MN, USA) and O3TM Regional Oximeter System ( We aimed to observe by doing it with O3 System, Masimo Corporation, Irvine, CA) devices.
Hepatic and renal tissue oxygenation | STO2 and O3 measurements at the end of the operation
  we will evaluate the effects of hepatic and renal StO2 measurement on early hypoperfusion and postoperative survival in hepatectomy cases, and peripheral tissue oxygen saturation measurement with StO2 InSpectra Tissue Spectrometer Model 1615 probe (Hutchinson Technology Inc. Hutchinson, MN, USA) and O3TM Regional Oximeter System ( We aimed to observe by doing it with O3 System, Masimo Corporation, Irvine, CA) devices.
Hepatic and renal tissue oxygenation | STO2 and O3 measurements at 24th hour postoperatively
  we will evaluate the effects of hepatic and renal StO2 measurement on early hypoperfusion and postoperative survival in hepatectomy cases, and peripheral tissue oxygen saturation measurement with StO2 InSpectra Tissue Spectrometer Model 1615 probe (Hutchinson Technology Inc. Hutchinson, MN, USA) and O3TM Regional Oximeter System ( We aimed to observe by doing it with O3 System, Masimo Corporation, Irvine, CA) devices.

SECONDARY OUTCOMES:
age | at 24th hour postoperatively
  If hepatic and renal StO2 measurement on early hypoperfusion will be affected by age, anatomical region, ASA physical condition, whether it will be affected by the vascular clamp duration and its correlation with the risk of developing postoperative complications.
ASA status | at 24th hour postoperatively
  If hepatic and renal StO2 measurement on early hypoperfusion will be affected by age, anatomical region, ASA physical condition, whether it will be affected by the vascular clamp duration and its correlation with the risk of developing postoperative complications.
Vascular clamp duration | İntraoperative duration of vascular clamp (minute)
  If hepatic and renal StO2 measurement on early hypoperfusion will be affected by age, anatomical region, ASA physical condition, whether it will be affected by the vascular clamp duration and its correlation with the risk of developing postoperative complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brazy JE, Lewis DV, Mitnick MH, Jobsis vander Vliet FF. Noninvasive monitoring of cerebral oxygenation in preterm infants: preliminary observations. Pediatrics. 1985 Feb;75(2):217-25. PMID 2982128
- [Background] Nardi O, Zavala E, Martin C, Nanas S, Scheeren T, Polito A, Borrat X, Annane D. Targeting skeletal muscle tissue oxygenation (StO2) in adults with severe sepsis and septic shock: a randomised controlled trial (OTO-StS Study). BMJ Open. 2018 Mar 19;8(3):e017581. doi: 10.1136/bmjopen-2017-017581. PMID 29555789